CLINICAL TRIAL: NCT06092086
Title: A Patient-Centric, Open-Label, Multicenter, Phase II Study of Lorlatinib Monotherapy in The First-Line Treatment of Patients With Advanced ALK-Positive Non-Small Cell Lung Cancer
Brief Title: Lorlatinib as the First-line Treatment in China Advanced ALK+ NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Principal Investigator, Yi-Long Wu, Principal Investigator, Guangdong Association of Clinical Trials
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTONG2203
Record Dates: First submitted 2023-07-21; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: ALK Positive Non-small Cell Lung Cancer
MeSH Terms: interventions — lorlatinib

STUDY DESIGN:
Intervention Model Description: Single drug administration
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CROWN Criteria (CC) Cohort、Compassionate use (CU) Cohort (Experimental)
  Interventions: Drug: Loratinib

INTERVENTIONS:
Drug: Loratinib — Continuous daily PO dosing of lorlatinib 100mg QD.
  Other Names: LORBRENA

SUMMARY:
This phase II study is aim to investigate the efficacy, resistance mechanism, safety profile of first-line lorlatinib in China advanced ALK+ non-small cell lung cancer (NSCLC). Participants will receive continuous daily PO dosing of lorlatinib 100mg QD.

DETAILED DESCRIPTION:
This is a patient-centric, two cohorts, open-label, multi-center, phase II study in China, designed to prospectively enroll 126 advanced ALK+NSCLC patients, including 84 subjects fulfilled CROWN criteria as "CROWN criteria (CC) cohort", and another 42 subjects beyond CROWN criteria as "compassionate use (CU) cohort". Subjects will receive continuous daily PO dosing of lorlatinib 100mg QD, from the date of first dosing until disease progression, unacceptable toxicity, or withdrawal for any reason, or death, whichever occurs first. The primary endpoints are progression-free survival (PFS) of CC cohort per investigator, and resistance mechanism of first-line lorlatinib. Secondary endpoints are 1/2/3-year PFS, cumulative rate of central nervous system (CNS) progression, intracranial-time to progression (IC-TTP), objective response rate (ORR) and intracranial ORR (IC-ORR), overall survival (OS), safety and PRO. Exploratory endpoints include evaluation of candidate biomarkers of sensitivity or resistance to lorlatinib, dynamic ctDNA change during treatment, and effective treatment after lorlatinib resistance.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria of CROWN Criteria (CC) Cohort

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:

1. Diagnosis:

   1. Study Population: Patients with histologically or cytologically confirmed diagnosis of locally advanced [(Stage IIIB/C not amenable for multimodality treatment) or metastatic (Stage IV) by American Joint Committee on Cancer (AJCC) v 7.0] ALK-positive NSCLC where ALK status is determined by the Ventana ALK (D5F3) Companion Diagnostic (CDx) IHC test performed on the Ventana ULTRA or XT Platforms, FISH, PCR, or next generation sequencing (NGS), or circulating tumor DNA (ctDNA).
   2. Tumor Requirements: At least 1 extracranial measurable target lesion per RECIST v. 1.1 that has not been previously irradiated. CNS metastases are allowed if asymptomatic and:

      1. Either untreated and not currently requiring corticosteroid treatment, or on a stable or decreasing dose of ≤10 mg QD prednisone or equivalent; or
      2. Local treatment has been completed with full recovery from the acute effects of radiation therapy or surgery prior to randomization, and if corticosteroid treatment for these metastases has been withdrawn for at least 4 weeks with neurological stability; or
      3. In case of leptomeningeal disease (LMD) or carcinomatous meningitis (CM) if visualized on magnetic resonance imaging (MRI), or if baseline CSF positive cytology is available.
   3. Tissue Requirements: All patients must have an archival formalin fixed, paraffin embedded (FFPE) tissue specimen available and collected prior to randomization. If archived tissue is unavailable, then a mandatory de novo biopsy must be performed.
2. No prior systemic NSCLC treatment for advanced (Stage IIIB/C not amenable for multimodality treatment) or metastatic (Stage IV) disease, including molecularly targeted agents (e.g., ALK TKIs), angiogenesis inhibitors, immunotherapy, or chemotherapy. Prior treatment for earlier Stages of the NSCLC only allowed if completed more than 12 months prior to randomization.
3. Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0, 1, or 2.
4. Age ≥18 years.
5. Adequate Bone Marrow Function, including:

   1. Absolute Neutrophil Count (ANC) ≥ 1,500/mm3 or ≥1.5 x 109/L;
   2. Platelets ≥100,000/mm3 or ≥100 x 109/L;
   3. Hemoglobin ≥9 g/dL.
6. Adequate Pancreatic Function, including:

   1. Serum total amylase ≤1.5 x upper limit of normal (ULN)*;
   2. Serum lipase ≤1.5 x ULN. *if total amylase >1.5 x ULN, but pancreatic amylase is within the ULN, then patient may be enrolled.
7. Adequate Renal Function, including:

   a. Serum creatinine ≤1.5 x ULN or estimated creatinine clearance ≥60 mL/min as calculated using the method standard for the institution.
8. Adequate Liver Function, including:

   1. Total serum bilirubin ≤1.5 x ULN;
   2. Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤2.5 x ULN (≤5.0 x ULN in case of liver metastases).
9. Acute effects of prior radiotherapy resolved to baseline severity or to CTCAE Grade ≤1 except for AEs that in the investigator's judgment do not constitute a safety risk for the patient.
10. Serum pregnancy test (for females of childbearing potential) negative at screening. Female patients of non-childbearing potential must meet at least 1 of the following criteria:

    1. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause (which may be confirmed with a serum follicle-stimulating hormone [FSH] level confirming the postmenopausal state if appropriate);
    2. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
    3. Have medically confirmed ovarian failure. All other female patients (including female patients with tubal ligations) are considered to be of childbearing potential.
11. Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.
12. Willing and able to comply with scheduled visits, treatment plans, laboratory tests and other procedures.

Inclusion Criteria of Compassionate use (CU) Cohort

1. Diagnosed as ALK-positive NSCLC as in CC cohort, but not fulfilled CC cohort inclusion criteria 2~9 as above mentioned.
2. No prior ALK TKI treatment for advanced (Stage IIIB/C not amenable for multimodality treatment) or metastatic (Stage IV) disease (e.g., alectinib, brigatinib).
3. Serum pregnancy test (for females of childbearing potential) negative at screening.
4. Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.
5. Willing and able to comply with scheduled visits, treatment plans, laboratory tests and other procedures.

Exclusion Criteria:

Subjects presenting with any of the following characteristics/conditions will not be included in this clinical study:

1. Spinal cord compression unless the patient has good pain control attained through therapy, and there is stabilization or recovery of neurological function for the 4 weeks prior to randomization.
2. Major surgery within 4 weeks prior to randomization. Minor surgical procedures (e.g., port insertion) are not excluded, but sufficient time should have passed for adequate wound healing.
3. Radiation therapy within 2 weeks prior to randomization, including stereotactic or partial brain irradiation. Patients who complete whole brain irradiation within 4 weeks prior to randomization or palliative radiation therapy outside of the CNS within 48 hours prior to randomization will also not be included in the study.
4. Gastrointestinal abnormalities, including inability to take oral medication; requirement for intravenous alimentation; prior surgical procedures affecting absorption including total gastric resection or lap band; active inflammatory gastrointestinal disease, chronic diarrhea, symptomatic diverticular disease; treatment for active peptic ulcer disease in the past 6 months; malabsorption syndromes.
5. Known prior or suspected severe hypersensitivity to study drugs or any component in their formulations.
6. Active and clinically significant bacterial, fungal, or viral infection including hepatitis B virus (HBV) or hepatitis C virus (HCV) (e.g., in case of known HBsAg or HCV antibody positivity), known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness.
7. Clinically significant vascular (both arterial and venous) and non-vascular cardiac conditions, (active or within 3 months prior to enrollment), which may include, but are not limited to:

   1. Arterial disease such as cerebral vascular accident/stroke (including Transient Ischemic Attack -TIA), myocardial infarction, unstable angina;
   2. Venous diseases such as cerebral venous thrombosis, symptomatic pulmonary embolism;
   3. Non-vascular cardiac disease such as congestive heart failure (New York Heart Association Classification Class ≥ II), second-degree or third-degree AV block (unless paced) or any AV block with PR >220 msec; or ongoing cardiac dysrhythmias of NCI CTCAE Grade ≥2, uncontrolled atrial fibrillation of any grade, bradycardia defined as <50 bpm (unless patient is otherwise healthy such as long-distance runners, etc.), machine-read Electrocardiogram (ECG) with QTc >470 msec, or congenital long QT syndrome.
8. Patients with predisposing characteristics for acute pancreatitis according to investigator judgment (e.g., uncontrolled hyperglycemia, current gallstone disease) in the last month prior to randomization.
9. History of extensive, disseminated, bilateral or presence of Grade 3 or 4 interstitial fibrosis or interstitial lung disease including a history of pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, interstitial lung disease, obliterative bronchiolitis, and pulmonary fibrosis.
10. Evidence of active malignancy (other than NSCLC, non-melanoma skin cancer, or localized prostate cancer or any in situ cancer which does not currently require treatment) within the last 3 years prior to randomization.
11. Concurrent use of any of the following food or drugs (consult the sponsor if in doubt whether a food or a drug falls into any of the above categories) within 12 days prior to the first dose of lorlatinib.

    1. Known strong CYP3A inhibitors (e.g., strong CYP3A inhibitors: grapefruit juice or grapefruit/grapefruit related citrus fruits [eg, Seville oranges, pomelos], boceprevir, cobicistat, conivaptan, itraconazole, ketoconazole, posaconazole, ritonavir alone and with danoprevir or elvitegravir or indinavir or lopinavir or paritaprevir or ombitasvir or dasabuvir or saquinavir or tipranavir, telaprevir, troleandomycin, and voriconazole. The topical use of these medications (if applicable), such as 2% ketoconazole cream, is allowed.
    2. Known CYP3A substrates with narrow therapeutic index, such as astemizole*, terfenadine*, cisapride*, pimozide, quinidine, tacrolimus, cyclosporine, sirolimus, alfentanil, fentanyl (including transdermal patch) or ergot alkaloids (ergotamine, dihydroergotamine) (*withdrawn from US market).
    3. Known strong CYP3A inducers (e.g., carbamazepine, enzalutamide, mitotane, phenytoin, rifampin, St. John's Wort). d. Known P-gp substrates with a narrow therapeutic index (e.g., digoxin).
12. Other severe acute or chronic medical or psychiatric condition, including recent (within the past year) or active suicidal ideation or behavior, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
13. Patients who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the Investigator, or patients who are Pfizer employees, including their family members, directly involved in the conduct of the study.
14. Participation in other studies involving investigational drug(s) within 2 weeks prior to study entry and/or during study participation.
15. Pregnant female patients; breastfeeding female patients; fertile male patients and female patients of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 97 days, if male or 35 days if female, after the last dose of investigational product under lorlatinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
PFS | From date of first dosing to first documented progression or death from any cause, whichever came first, assessed up to 3 years.
  Progression Free Survival (PFS) is defined as the time from start of lorlatinib treatment to the date of disease progression as defined by RECIST v1.1 per investigator review or death due to any cause, whichever occurred first.
Resistance mechanism of lorlatinib | From date of first dosing to first documented progression or death from any cause, whichever came first, assessed up to 3 years.
  Resistance mechanism of first-line lorlatinib treatment by tumor tissue, and peripheral blood ctDNA (circulating tumor Deoxyribonucleic acid) biomarkers including, but not limited to, ALK gene rearrangement and/or ALK kinase domain mutations as measured by next-generation sequencing (NGS);

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Long Wu, MD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial Perople's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin JX, Zhou Q, Yan HH, Liu AW, Wu GW, Chu Q, Du YY, Cui JW, Cheng Y, Yang Y, Xu HP, Tu HY, Wu YL, Liu SM. A Patient-Centric, Open-Label, Multicenter, Phase II Study of Lorlatinib Monotherapy in the First-Line Treatment of Patients With locally Advanced or Metastatic ALK-Positive Non-Small Cell Lung Cancer (CTONG2203). Clin Lung Cancer. 2025 Sep;26(6):515-519. doi: 10.1016/j.cllc.2025.05.014. Epub 2025 May 28. PMID 40541556